CLINICAL TRIAL: NCT05566418
Title: Immediate and Long Term Effects of Mulligan Mobilization With and Without Myofascial Release on Pain, Grip Strength and Function in Patients With Lateral Epicondylitis
Brief Title: Immediate and Longterm Effects of Mulligan Mobilization With and Without Myofascial Release on Pain,Grip Strength and Function in Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 898
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Ultrasonic Therapy; Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Parallel designed randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: This study will be single blinded. Patients will be assessed by a senior Physiotherapist then divided into two groups for treatments. The assessor will be unaware of the treatment given to both groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): Group A will get standard therapy and the Mulligan mobilization technique for 12 sessions. A Mulligan mobilization belt will be wrapped around the subject's proximal forearm, close to the elbow joint line, and then wrapped around the therapist's shoulder. This will be done with the therapist's other hand on the distal humerus. The belt will give the subject's forearm a 10-to 15-second lateral glide. The patient will be instructed to constantly extend their wrists while the therapist applies manual resistance to their attempts, and the therapist will continue to work on the patient. When the user can fully extend their wrist without discomfort, the lateral glide will be abolished. Three repeats will be performed, each separated by a fifteen-to twenty-second interval.
- Group B (Experimental): In addition to the standard treatment, Group B participants will receive 12 sessions of myofascial release technique and Mulligan mobilization. Participants will be instructed to lie supine on the plinth with the afflicted arm internally rotated, elbow slightly flexed and pronated, and palm of hand on the plinth. While standing on the side of the body affected by the ailment being treated, the therapist turned their body to face the affected hand. Myofascial release will be performed on the patient The therapeutic session will last five minutes and will be repeated twice.
  Interventions: Other: mulligan mobilization; Other: myofascial release

INTERVENTIONS:
Other: mulligan mobilization — Mulligan mobilization belt will be wrapped around the subject's proximal forearm, close to the elbow joint line, and then wrapped around the therapist's shoulder. This will be done with the therapist's other hand on the distal humerus. The belt will give the subject's forearm a 10-to 15-second lateral glide.
  Other Names: transcutaneous electric nerve stimulation,Cryo-therapy, Ultrasonic therapy, strengthening exercises
  Arms: Group B
Other: myofascial release — Myofascial release will be performed on the patient, commencing at the common extensor origin and progressing all the way to the extensor retinaculum in the wrist. The periosteum will be engaged with the fingertips, with contact progressing inferiorly to the common extensor tendon and then to the wrist's extensor retinaculum
  Arms: Group B

SUMMARY:
This study will help to determine the immediate and long term effects of Mulligan mobilization with and without myofascial release on pain, grip strength and function in patients with lateral epicondylitis

DETAILED DESCRIPTION:
Tennis elbow patients usually experience diminished grip strength, decreased functional activities, and increased pain, all of which can have a significant impact on everyday activities. Tennis elbow can also be caused by excessive elbow use. The following is a description of the basic clinical manifestation of tennis elbow, as well as the most commonly reported symptoms of people suffering from the condition: Tennis elbow is easily identified and confirmed with a test that produces discomfort, palpable tenderness over the lateral epicondyle facet, resisted wrist extension, resisted middle finger extension, and passive wrist flexion. Tennis elbow is a common elbow disease caused by excessive use. Furthermore, despite some difficulty, the patient must be able to extend his or her wrist and middle finger. The goal of this study is to find out how Mulligan Mobilization with and without myofascial release affects pain, grip strength, and function in people with lateral epicondylitis in the short and long term.

Mulligan mobilisation and myofascial release have both been shown to be effective treatments for lateral epicondylitis. The purpose of this study is to look into the short-and long-term advantages of myofascial release and Mulligan mobilisation. No research has been conducted to evaluate whether mulligan mobilisation with or without myofascial release benefits people with lateral epicondylitis in terms of pain, grip strength, and overall function. This study will not only help therapists come up with treatment goals for lateral epicondylitis, also known as tennis elbow, but it will also add credibility to the existing body of literature.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 20 years to 40 years ,both males and females
2. Diagnosed cases of lateral epicondylitis by senior physiotherapist
3. Acute and sub-acute cases
4. Numeric Pain Rating Scale 4 and above
5. Positive cozen test, Mills test, middle finger extension test

Exclusion Criteria:

* H/o

  1. Active medications.
  2. Dermatitis, malignancy or hazardous to myofascial release.
  3. Recent trauma, fracture
  4. Prior surgeries of elbow, tendon ruptures
  5. Any Neurological conditions like nerve compression
  6. Swelling around the elbow joint

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
change from baseline in pain at week 4th | baseline and 4th week
  Numeric pain rating scale will be used to assess the pain level. A score of 0 means there is no pain, while a score of 10 means the worst pain

OTHER OUTCOMES:
change from baseline in grip strength at week 4th | baseline and 4th week
  A handheld dynamometer will be used to assess the maximal grip strength.
change from baseline in functional ability at week 4th | baseline and 4th week
  The Patient-Rated Tennis Elbow Evaluation (PRTEE) is a strong, dependable, and sensitive outcome measure used to identify functional activity participation issues. It consists of 15 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Sumra Riaz, MS-PTM, Study Director — University of Lahore
Locations (1):
- Sumra Riaz, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No